CLINICAL TRIAL: NCT00736294
Title: Prevention of Atrial Fibrillation by the Prescription of Inhibition Conversion Enzyme (ICE) After Radiofrequency Ablation of Atrial Flutter
Brief Title: Prevention of Atrial Fibrillation by Inhibition Conversion Enzyme (ICE) After Radiofrequency Ablation of Atrial Flutter
Acronym: PREFACE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Difficulty to include patients
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Sanofi (Industry); Ministry of Health, France (Other Government); LivaNova (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0608066; 2006-007032-10 (Other: ANSM)
Record Dates: First submitted 2008-08-14; First posted 2008-08-15 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Atrial Fibrillation; Atrial Flutter
Keywords: Catheter Ablation, Radiofrequency; Angiotensin-Converting Enzyme Inhibitors
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter | interventions — Ramipril

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ramipril (Experimental): Inhibition Conversion Enzyme
  Interventions: Drug: Ramipril
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ramipril — 5 mg/d from D1 to M3 10 mg/d from M3 to M12 Tablets
  Arms: Ramipril
Drug: Placebo — 5 mg/d from D1 to M3 10 mg/d from M3 to M12 Tablets
  Arms: Placebo

SUMMARY:
Atrial Flutter [AFL] is a relatively frequent arrhythmia, considered as benign, but associated with both invalidating symptoms and thromboembolic risk. The objective of the treatment consists to on the one hand the sinus rhythm [SR] restoration and on the other hand the prevention of the long-term recurrence. In this clinical setting, AFL radiofrequency ablation [RFA] became the first line therapy due to its both high effectiveness and safety. The effectiveness of AFL RFA is attenuated by the subsequent risk of atrial fibrillation [AFib] close to 25% at 1 year. This risk of subsequent AFib is related to the common substrate between both arrhythmias.

When AFib occurs, the interest to maintain the SR is still required, even if recent studies did not show a significant difference in term of total mortality between rate or rhythm control strategies [AFFIRM, RACE and PIAF studies]. The studies published underlined the anti-arrhythmic drugs limits in patients with both arrhythmias [AFib and AFL]. After years centered on the mechanisms and the electric treatments of AFib, researchers are nowadays focusing on the study's evaluation of the atrial tissue substrate.

Accordingly, the renin-angiotensin system role was investigated in many works. Indeed, angiotensin II plays a role in the modification of atrial pressure and in the fibers stretching ["stretch"], conditions required for the development of AFib. Angiotensin II is also a factor implied in the tissue fibrosis leading to tissue proliferation and collagen alteration. These mechanisms lead to atria cells conduction disorders and refractory periods modification. Moreover, the enzyme of conversion expression and the angiotensin II receptors deterioration were observed in patients with AFib.

This brings to the concept of AFib treatment while interfering on tissue remodeling by the way of renin-angiotensin system. Drugs such as the angiotensin converting enzyme inhibition [ACEI] may reduce AFib in patients with heart failure. No randomized study so far has compared the ACEI drugs against placebo among high-risk patients of AFib in post AFL RFA area. On the basis of experimental and clinical study, the investigators seek to evaluate the ACEI use in the prevention of AFib in an AFL post RFA ablation.

DETAILED DESCRIPTION:
The main goal of this study is to compare within 12 months, the effectiveness of an ACEI [Ramipril] versus placebo on the prevention of AFib after AFL RFA.

This study is a randomized, prospective, double blind, multicenter study comparing ramipril vs. placebo in 2 parallel groups.

ELIGIBILITY:
Inclusion Criteria:

* first atrial flutter, or recurrence of atrial flutter
* affiliated or a beneficiary of a social security category
* treated by radiofrequency ablation (< 72 h)
* having signed the inform consent form

Exclusion Criteria:

* contra-indication to right catheterism
* contra-indication to angiotensin converting enzym inhibitors
* contra-indication to anticoagulation treatment
* having already a angiotensin converting enzym inhibitor treatment
* recent (< 3 months) hearth failure with left ventricular ejection fraction < 45%
* pregnant women or breast-feeding
* severe renal disease
* serum potassium > 5 mmol/l
* requiring a antiarrythmic treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2008-07; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
At least one relevant symptomatic or asymptomatic atrial fibrillation event | From D1 to M12

SECONDARY OUTCOMES:
All relevant cardiovascular event | From D1 to M12
Secondary effects of the treatment | From D1 to M12

CONTACTS AND LOCATIONS:
Overall Officials: Antoine DA COSTA, PhD MD, Principal Investigator — CHU de Saint-Etienne
Locations (8):
- France (8):
  - CHU de Brest, Brest
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - CHU de Grenoble, Grenoble
  - CHU de Montpellier, Montpellier
  - Polyclinique des Fleurs, Ollioules
  - CHU de Rennes, Rennes
  - CHU de Rouen, Rouen
  - CHU de Saint-Etienne, Saint-Etienne

REFERENCES:
- [Background] Da Costa A, Thevenin J, Roche F, Romeyer-Bouchard C, Abdellaoui L, Messier M, Denis L, Faure E, Gonthier R, Kruszynski G, Pages JM, Bonijoly S, Lamaison D, Defaye P, Barthelemy JC, Gouttard T, Isaaz K; Loire-Ardeche-Drome-Isere-Puy-de-Dome Trial of Atrial Flutter Investigators. Results from the Loire-Ardeche-Drome-Isere-Puy-de-Dome (LADIP) trial on atrial flutter, a multicentric prospective randomized study comparing amiodarone and radiofrequency ablation after the first episode of symptomatic atrial flutter. Circulation. 2006 Oct 17;114(16):1676-81. doi: 10.1161/CIRCULATIONAHA.106.638395. Epub 2006 Oct 9. PMID 17030680
- [Background] Da Costa A, Romeyer-Bouchard C, Zarqane-Sliman N, Messier M, Samuel B, Kihel A, Faure E, Isaaz K. Impact of first line radiofrequency ablation in patients with lone atrial flutter on the long term risk of subsequent atrial fibrillation. Heart. 2005 Jan;91(1):97-8. doi: 10.1136/hrt.2003.033308. No abstract available. PMID 15604348
- [Background] Madrid AH, Peng J, Zamora J, Marin I, Bernal E, Escobar C, Munos-Tinoco C, Rebollo JM, Moro C. The role of angiotensin receptor blockers and/or angiotensin converting enzyme inhibitors in the prevention of atrial fibrillation in patients with cardiovascular diseases: meta-analysis of randomized controlled clinical trials. Pacing Clin Electrophysiol. 2004 Oct;27(10):1405-10. doi: 10.1111/j.1540-8159.2004.00645.x. PMID 15511250
- [Background] Heart Outcomes Prevention Evaluation Study Investigators; Yusuf S, Sleight P, Pogue J, Bosch J, Davies R, Dagenais G. Effects of an angiotensin-converting-enzyme inhibitor, ramipril, on cardiovascular events in high-risk patients. N Engl J Med. 2000 Jan 20;342(3):145-53. doi: 10.1056/NEJM200001203420301. PMID 10639539